CLINICAL TRIAL: NCT04666376
Title: Vitrified Ovarian Tissue in Cancer Patients: Assessing the Technique in Vietnam
Brief Title: Assessing the Technique of Ovarian Tissue Cryopreservation by Vitrification in Vietnam
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Mỹ Đức Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 15/20/DD-BVMD
Record Dates: First submitted 2020-11-30; First posted 2020-12-14 (Actual); Last update posted 2020-12-17 (Actual); Status verified 2020-11

CONDITIONS: Ovarian Tissue Cryopreservation; Vitrification

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Vitrified ovarian tissue (Other): Ovarian tissue will be vitrified and warmed by Ova kit type M protocol.
  Interventions: Other: evaluation of the effectiveness of vitrification technique on ovarian tissue quality

INTERVENTIONS:
Other: evaluation of the effectiveness of vitrification technique on ovarian tissue quality — there are 3 types of experiments in each group, including Follicle survival evaluation by Neutral red staining, Histological evaluation by Hematoxylin and Eosin staining, 2.4. Evaluation GDF-9 and Caspase-3 gene expression by real-time PCR.

SUMMARY:
Ovarian tissue cryopreservation (OTC) is a new approach on fertility preservation for young female patients with cancer. It is now used by many IVF centers in the world. However, this is the first study which OTC by vitrification is carried on and assessed the effectiveness of the technique.

DETAILED DESCRIPTION:
Ovaries from all less than 45 year-old breast cancer patients who undergo oophorectomy by laparoscopy after treated with chemotherapy will be enrolled to the study. Pieces of cortex of each patient will divide into two groups. Group 1 is fresh fragments (control group) and group 2 is vitrified group. Ovarian tissues in group 2 will be vitrified or warmed with medium and devices of Ova-kit type M (Kitazato, Japan).

Cortex fragments of each group will have:

* Follicle survival evaluation by Neutral red staining
* Histological evaluation by Hematoxylin and Eosin staining
* Evaluation relative Growth Differentiation Factor 9 (GDF-9) and Caspase-3 gene expression by real-time Polymerase chain reaction (PCR).

Comparison of data collected from 2 groups will be carried on to evaluate the effectiveness of the technique before applying this technique for cancer patients in Vietnam.

ELIGIBILITY:
Inclusion Criteria:

* Ovaries from all less than 45 year-old breast cancer patients who undergo oophorectomy by laparoscopy after treated with chemotherapy

Exclusion Criteria:

* The volume of ovaries is less than 2/3 of normal 3cm (L) x 2.5cm (H) x 1.5cm (W) ovary.

Max Age: 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 43 (Estimated)
Dates: Start 2021-01-01 (Estimated); Primary Completion 2021-02-01 (Estimated); Study Completion 2022-01-31 (Estimated)

PRIMARY OUTCOMES:
Rate of Survivable follicle | After 4 hours stained by Neutral red
  Percentage of survivable follicles per counted follicles in one fragment

SECONDARY OUTCOMES:
Rate of Healthy follicle by histological analysis | Immediately after tissue stained by Hematoxylin and Eosin
  Healthy follicles of primordial, primary, secondary follicles will be counted in one slide
The relative expression ratio ( R ) of genes in follicles | Immediately after the intervention
  Follicles in ovarian tissue will be collected, complementary deoxyribonucleic acid (cDNA) synthesis after messenger ribonucleic acid (mRNA) purification, relative quantification PCR for detecting gene expression

CONTACTS AND LOCATIONS:
Overall Officials: Tuong M Ho, MD, MCE, Principal Investigator — Hope Research Center
Locations (1):
- My Duc Hospital, Ho Chi Minh City, Vietnam